CLINICAL TRIAL: NCT02775058
Title: Clinical Evaluation Protocol Post Market Follow Up Pavia CP009 SYNERGOSS PXX Observational
Brief Title: CP009 SYNERGOSS PXX Observational
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nobil Bio Ricerche srl (Industry)
Responsible Party: Sponsor
Other Study IDs: CP009
Record Dates: First submitted 2016-03-24; First posted 2016-05-17 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-06

CONDITIONS: Mouth, Edentulous
MeSH Terms: conditions — Mouth, Edentulous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — vital bone specimen sampled during surgery for dental implant placement
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- patients: The subjects enrolled in this CI just received dental grafting by the device under evaluation and in any case will be subject to the same procedures foreseen for this CI for the dental implant surgery.
  Interventions: Device: synergoss Pxx

INTERVENTIONS:
Device: synergoss Pxx — dental grafting

SUMMARY:
The device under investigation is SYNERGOSS, a CE (European Community CE) marked device.

Synergoss is a granulated bone graft intended for use in dental applications. It is composed of a ceramic composite of Hydroxihapatite and Tricalciumphosphate in granules, coated with a dedicated collagen coating (porcine origin), obtained by means of collagen crosslinking on the ceramic granule surface.

The purpose of the study is to confirm the foreseen efficacy and tolerability of SYNERGOSS, a synthetic dental graft coated with collagen. For this observational study, we will enroll patients that already received a surgical intervention for sinus augmentation/ socket preservation by means of SYNERGOSS to maintain and regenerate bone before installation of endosseous titanium implants to support a fixed prosthesis. Patients will be enrolled just before they receive the surgery for the installation of endosseous titanium implants, about 24 weeks after the first surgery for the implant of SYNERGOSS.

The primary hypothesis is to demonstrate that SYNERGOSS consistently obtains the foreseen clinical benefit as declared in the Technical File.

The secondary hypothesis is to demonstrate that SYNERGOSS side effects and risks match those declared in the Technical File.

The study design is a

* National
* Monocentric
* Prospective: the participants are identified and then followed forward in time.
* Observational: participants that have recently received the grafting with SYNERGIES as part of normal and foreseen clinical procedures are enrolled in the study when they receive surgery for titanium implant placement and observed over time, with no substantial intervention other than the foreseen clinical treatment

ELIGIBILITY:
Inclusion Criteria:

* • Received in the past 16-24 weeks a bone graft for sinus lift or socket preservation with the ID

  * Capable of giving a valid informed consent
  * ASA 1, ASA 2
  * agrees to return for follow-up visits up to 2 years

Exclusion Criteria:

* • Uncontrolled Diabetes

  * Patients with psychiatric diseases
  * Neoplasic, immunodepressive, renal or liver major illnesses
  * Local radiotherapy
  * Major bruxism or major differences in the maxilla or mandubilar area
  * Drug or alcohol abuse
  * Major bone metabolism disorders
  * Heavy smokers (more than 10/day)
  * bisphosphonate treatment of major ostheoporosys or bone neoplasia
  * Pregnant women
  * Sinus illnesses
  * Contraindications to implant supported prostheses
  * Patients ASA 3,ASA 4, ASA5
  * Surgical intervention contraindications

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects enrolled in this CI just received dental grafting and in any case will be subject to the same procedures foreseen for this CI for the dental implant surgery.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
• Bone Volume total (%BV) | 4-6 months
  The specimen, extracted from the bone of the patient, will be evaluated to define the quantity of total bone volume as compared to the specimen volume
• graft Volume (%graft) | 4-6 months
  The specimen, extracted from the bone of the patient, will be evaluated to define the quantity of residual, non absorbed graft volume as compared to the specimen volume
• vital bone (%VB). | 4-6 months
  The specimen, extracted from the bone of the patient, will be evaluated to define the quantity of vital, new formed bone volume as compared to the specimen volume
• device radiologic density (in a qualitative scale ranging from 1 to 4) | 4-6 months
  the radiological density is visually evaluated by the investigator

CONTACTS AND LOCATIONS:
Overall Officials: Ruggero Rodriguez y Baena, Principal Investigator — POLICLINICO S. MATTEO - PAVIA
Locations (1):
- Policlinico S. Matteo - Pavia, Pavia, PV, Italy